CLINICAL TRIAL: NCT02130960
Title: Resting Metabolic Rate Reliability
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC027
Record Dates: First submitted 2014-04-30; First posted 2014-05-06 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Resting Metabolic Rate Reliability
Keywords: RMR; Reliability; Obese; Energy Expenditure; Resting Energy Expenditure; Resting Metabolic Rate
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This research is being conducted to study the reliability of a method used to measure resting metabolic rate, or how much energy a person expends while at rest.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years old
* BMI of 19 - 40 kg/m2
* Women must not be pregnant or planning to become pregnant

Exclusion Criteria:

* Age less than 18 or greater than 65
* BMI less than 19 or greater than 40
* Tobacco use
* Taking medications that affect metabolic rate (unless weight stable for past 3 months)
* Any disease that affects the metabolic rate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include up to 15 men and 15 women age 18 -65 years old with a BMI of 19 - 40 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Resting Metabolic Rate by Indirect Calorimetry | At least 3 days
  The within-subject coefficient of variation for resting metabolic rate (RMR) will be less than 10%. Testing will occur on non-consecutive days, with a compliance and menstrual cycle questionnaire prior to testing.

SECONDARY OUTCOMES:
Respiratory Quotient Variation | At least 3 days
  The within-subject coefficient of variation for respiratory quotient (RQ) will be less than 10%. Testing will occur on non-consecutive days, with a compliance and menstrual cycle questionnaire prior to testing.
Sense Wear Mini Armband verses Indirect Calorimetry | At least 3 days
  The limits of agreement of Sense Wear Mini Armband (SWA)-estimated resting energy expenditure (REE) with indirect calorimetry measures of REE will be large (+ 500 kcal). Testing will occur on non-consecutive days, with a compliance and menstrual cycle questionnaire prior to testing.

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States